CLINICAL TRIAL: NCT05080608
Title: Patients´ Experiences of Changed Physical Activity Level Following Nerve Injury in the Upper Limb- a Qualitative Study
Brief Title: Nerve Injury in the Hand, an Interview Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Karolinska Institutet (Other)
Collaborators: Department of Hand surgery Södersjukhuset (Other)
Responsible Party: Principal Investigator, Cecilia Mellstrand Navarro, Principal Investigator, Karolinska Institutet
Other Study IDs: Nerve injury interview
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Nerve Injury
MeSH Terms: interventions — Surgical Procedures, Operative; Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nerve injury: This is an interview study of patients with injury to the median, ulnar or digital nerve or brachial plexus injury.
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — Treatment according to clinical practise
  Other Names: Rehabilitation

SUMMARY:
This qualitative study sought to explore the exerience of change in physical activity due to nerve injury in the arm and hand.

DETAILED DESCRIPTION:
Aim:

Has the physical activity level changed in connection with the nerve injury. Experiences of factors influensing this change.

Population: Patients surgically treated for digital,median,ulnar-or plexus nerveinjuries at Södersjukhuset or Universitets sjukhuset in Linköping. 1-3 years ago. Age 18-75.

Method: Interviews are carried out over the phone, digitally recorded and trascribed. The analysis is inductive approach.

ELIGIBILITY:
Inclusion Criteria:

* Injury to the median, ulnar or digital nerve or injury to the brachial plexus.
* 1-5 years post injury.

Exclusion Criteria:

* Severe psychiatric disease.
* Drug or alcohol abuse.
* Insufficient language understanding.
* Severe diabetes mellitus with nerve complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated surgically due to Injury to the median, ulnar or digital nerve or injury to the brachial plexus. 1-5 years post injury.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Interview | 1-5 years post injury
  A semi structured interview will be conducted, utilizing semi structured interview. Themes regarding changes in physical activity related to the nerve injury will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Arner, Professor, Study Director — Karolinska Institutet; Cecilia Mellstrand Navarro, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet södersjukhuset, Stockholm, Sweden